CLINICAL TRIAL: NCT07057245
Title: Effects of Daily Protein Supplementation on Brain Function in Older Adults With Overweight or Obesity
Brief Title: Effects of Protein Supplementation on Brain Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Cosun (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 24-053
Record Dates: First submitted 2025-05-02; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Brain Vascular Function; Cognitive Function; Satiety; Cerebral Blood Flow; Brain Insulin Sensitivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plant-based protein (Experimental)
  Interventions: Dietary Supplement: Protein supplementation with a plant-based protein isolate
- Animal-based protein (Experimental)
  Interventions: Dietary Supplement: Protein supplementation with an animal-based protein isolate
- Control arm (Other): Cornstarch providing no extra protein
  Interventions: Other: Control arm - cornstarch

INTERVENTIONS:
Dietary Supplement: Protein supplementation with an animal-based protein isolate — Study participants will consume, in random order, twice daily (2 x ~20 g) a plant protein (fava bean protein isolate), animal protein (milk protein isolate) or control (cornstarch providing no extra protein)
  Arms: Animal-based protein
Dietary Supplement: Protein supplementation with a plant-based protein isolate — Study participants will consume, in random order, twice daily (2 x ~20 g) a plant protein (fava bean protein isolate), animal protein (milk protein isolate) or control (cornstarch providing no extra protein)
  Arms: Plant-based protein
Other: Control arm - cornstarch — Study participants will consume, in random order, twice daily (2 x ~20 g) a plant protein (fava bean protein isolate), animal protein (milk protein isolate) or control (cornstarch providing no extra protein)
  Arms: Control arm

SUMMARY:
Protein-rich foods may improve brain insulin-sensitivity, which is important for cognitive and metabolic health, and may also translate into an improved food intake regulation. It is therefore pertinent to delineate the effects of plant-derived proteins, which are a more sustainable alternative to animal-derived proteins, on brain insulin-sensitivity and related functional benefits. The hypothesis is that daily plant-derived or animal-derived protein supplementation improves brain vascular function and insulin-sensitivity, thereby improving cognitive performance and appetite control in overweight or obese older men and women.

The primary objective is to investigate in overweight or obese older adults the effect of daily protein supplementation for two weeks with either a plant-derived protein or an animal-derived protein on vascular function and insulin-sensitivity in the brain, while changes in cognitive performance and appetite-related brain reward activity will also be evaluated (secondary study objectives). Cerebral blood flow responses before (brain vascular function) and after the administration of intranasal insulin spray (brain insulin-sensitivity) will be quantified by the gold standard magnetic resonance imaging (MRI)-perfusion method Arterial Spin Labeling (ASL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 60-75 years (older adults)
* BMI between 25-35 kg/m2 (overweight or obese)
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Intolerant to milk products or fava bean allergy
* Vegetarians
* Left-handedness
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of products or dietary supplements known to interfere with the main outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid, or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases, and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging (e.g., pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow responses before (brain vascular function) and after the administration of intranasal insulin spray (brain insulin-sensitivity) | Measured after 2 weeks of supplementation with protein isolate or control

SECONDARY OUTCOMES:
Cognitive performance | Measured after 2 weeks of supplementation with protein isolate or control
  Cognitive performance will be assessed with a neuropsychological test battery
Appetite-related brain reward activity | Measured after 2 weeks of supplementation with protein isolate or control
  Blood oxygenation level-dependent (BOLD)-functional MRI (fMRI) response to food cues

OTHER OUTCOMES:
Transcranial Doppler ultrasound | Measured after 2 weeks of supplementation with protein isolate or control
  Blood flow velocity in the MCA
Blood pressure | Measured at baseline and after two weeks of supplementation with protein isolate or control
  Office BP (SBP and DBP) measured in mmHg
Heart rate | Measured at baseline and after two weeks of supplementation with protein isolate or control
  Heart rate (HR) measured in beats/min
Metabolic risk markers - Fasting lipids | Measured at baseline and after two weeks of supplementation with protein isolate or control
  Fasting lipids:
  * Fasting serum triacylglycerol (TAG) concentrations in mmol/L will be measured
  * Fasting serum total cholesterol (TC) and HDL-C in mmol/L will be measured
Metabolic risk markers - glucose and insulin | Measured at baseline and after two weeks of supplementation with protein isolate or control
  Fasting glucose and insulin:
  * Fasting plasma glucose concentrations in mmol/L will be measured
  * Fasting serum insulin concentrations in mmol/L will be measured
Metabolic risk markers - Low-grade systemic inflammation and microvascular function | Measured at baseline and after two weeks of supplementation with protein isolate or control
  Low-grade systemic inflammation and microvascular function:
  * Fasting hemostatic factors and plasma markers related to systemic inflammation will be measured to assess low-grade systemic inflammatory responses (e.g. CRP)
  * Fasting plasma markers related to microvascular function will be measured to determine microvascular responses
Single nucleotide polymorphisms (SNPs) | Measured once during the start of the study
  Leucocytes will be isolated from EDTA blood. DNA will be isolated from these leucocytes according to standard procedures. DNA will be used for analyzing the presence of known SNPs in genes encoding proteins known to play a role in cholesterol metabolism.
Perceived hunger and satiety | Measured after 2 weeks of supplementation with protein isolate or control
  Visual analogue scale (VAS) questionnaires will be used to assess perceived feelings of hunger, fullness, desire to eat, and prospective food consumption.
Anthropometric measurements | Measured at baseline and after two weeks of supplementation with protein isolate or control
  At all test days, anthropometric measurements (weight, length, waist and hip circumferences as indirect measures of fat distribution, and skinfold measurements) will be measured
Dietary intake | Measured after 2 weeks of supplementation with protein isolate or control
  At the end of both interventions, food intake will be measured using a validated food frequency questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands